CLINICAL TRIAL: NCT06122870
Title: Double-blind, Placebo-Controlled Trial Assessing the Efficacy and Safety of CampETEC Hyperimmune Bovine Colostrum (HBC) for the Prevention of Campylobacter-Mediated Diarrheal Diseases
Brief Title: CampETEC Hyperimmune Bovine Colostrum (HBC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); The Henry M. Jackson Foundation for the Advancement of Military Medicine, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIR 360; IRB00026228 (Other: JHSPH IRB)
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteer
Keywords: Campylobacter; CG8421; Challenge; Hyperimmune Bovine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CampETEC HBC group (Experimental): CampETEC HBC (hyper immune bovine colostrum) and challenge strain C. jejuni CG8421
  Interventions: Biological: CampETEC HBC product; Biological: C. jejuni CG8421 Challenge strain
- Placebo ProMilk 85 group (Placebo Comparator): ProMilk 85 (placebo) and challenge strain C.jejuni CG8421
  Interventions: Biological: ProMilk 85; Biological: C. jejuni CG8421 Challenge strain

INTERVENTIONS:
Biological: CampETEC HBC product — Immunoglobulin from bovine milk/colostrum and challenge strain
  Arms: CampETEC HBC group
Biological: ProMilk 85 — Placebo ProMilk 85
  Arms: Placebo ProMilk 85 group
Biological: C. jejuni CG8421 Challenge strain — Challenge strain C. jejuni CG8421

SUMMARY:
Gastrointestinal infections cause significant morbidity in the form of acute diarrheal illness in the United States (US) and among travelers to low- and middle-income countries (LMICs). One approach is to use passive protection (antibodies) to prevent infection. The purpose of this study are to assess the safety and tolerability of serum-derived bovine immunoglobulins in healthy adult subjects when orally administered and to estimate protective efficacy of those preparations against moderate-severe diarrhea upon challenge with Campylobacter C. jejuni strain CG8421.

DETAILED DESCRIPTION:
Controlled Human Infection ModelCampylobacter is a leading cause of foodborne disease in the US, is associated with 7.5 million disability adjusted life years globally and is a pathogen of concern in pediatric populations in LMICs and adult travelers to those same regions. Campylobacteriosis disproportionately affects poor and marginalized populations of the developing world and is particularly hazardous to the health and viability of infants in this region. The global diarrhea burden caused by Campylobacter spp. is estimated to include 88 million episodes in children aged ≤5 years, resulting in roughly 41,000 deaths. Among all age groups, the estimates of episodes and deaths are roughly 172 million and 75,000, respectively. In the US, Campylobacter causes more than 1.5 million illnesses each year mostly due to the handling and consumption of raw or undercooked poultry. For travelers, Campylobacter causes a severe form of Traveler's Diarrhea (TD), often associated with longer illness duration, increased number of unformed stools, and a high frequency of other symptoms (abdominal pain, nausea, vomiting, and fever) in comparison with other TD etiologies. In addition, Campylobacter infection is associated with several important sequelae, including Guillain-Barré syndrome (GBS), reactive arthritis, irritable bowel syndrome, and, to a lesser extent, inflammatory bowel disease. Until recently, campylobacteriosis has been viewed as a self-limiting illness that is ameliorated by antibiotic treatment; however, resistance of Campylobacter to antibiotics, particularly fluoroquinolones, has become a concern. Thus, alternative measures to control infection are needed. C. jejuni lacks virulence factors analogous to those of better-characterized pathogens. However, the C. jejuni Capsular polysaccharide (CPS) was recently identified and is now recognized as a major virulence factor and the focus of vaccine development efforts. A total of 47 C. jejuni capsule types have been described and through structure homology can be collapsed into 35 groups. Based on scant epidemiological data from developing countries, it appears that a limited number of C. jejuni capsule types are responsible for the majority of the disease.

One modality that has shown considerable promise in diarrhea prevention is passive, oral administration of HBC, hyperimmune bovine colostrum. In a number of clinical trials, HBC as well as bovine serum IgG (BSIgG), with specific activity against enteropathogens like Enterotoxigenic E. coli (ETEC), Shigella, and rotavirus, have shown to prevent diarrheal disease in Controlled Human Infection Models (CHIM). This study will establish the foundation for evaluating HBC products against Campylobacter.

This randomized, double-blinded, placebo- controlled study will explore if Hyperimmune bovine colostrum provides protection against oral challenges with Campylobacter in healthy adult participants. There will be an inpatient admission of approximately 30 subjects. Participants will be randomized to receive the investigational product (IP) or placebo three times daily following meals beginning 2 days prior to challenge. Each volunteer will be challenged with C.jeuni strain CG8421 on Day 1. The investigational product/placebo will be administered for a total of 7 days, or until antibiotic treatment has been administered. The investigators hypothesize that HBC will provide protection against C. jejuni strain CG8421 mediated moderate to severe diarrhea upon challenge.

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18 and 50 years of age, inclusive.
* General good health, without significant medical illness, abnormal physical examination findings, or clinical laboratory abnormalities, as determined by principal investigator (PI) or PI in consultation with the research monitor and sponsor.
* Demonstrate comprehension of the protocol procedures, requirements, and CHIM by passing a written examination (passing grade ≥ 70%).
* Willing to participate, as evidenced by signing the informed consent document.
* Available for all planned follow-up visits.
* Negative serum pregnancy test at screening and negative serum and/or urine pregnancy test on the day of admittance to the inpatient phase for participants of childbearing potential. Participants of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence from intercourse with a male partner is acceptable. Participants who no longer have childbearing potential must have this documented (e.g., tubal ligation or hysterectomy).

Exclusion Criteria:

General health issues

* Presence of a significant medical condition (e.g., psychiatric conditions such as significant anxiety, depression, or somatization disorder; gastrointestinal disease, such as peptic ulcer, symptoms or evidence of active gastritis/dyspepsia, gastroesophageal reflux disease, inflammatory bowel disease, irritable bowel syndrome (as suggested by the functional bowel disorder survey or medical diagnosis); alcohol or illicit drug abuse/dependency; or laboratory abnormalities that in the opinion of the investigator preclude participation in the study. Significant medical conditions include HIV, active Hepatitis B or C infection, ongoing immunosuppression for any reason, autoimmune disease, evidence of cardiac, pulmonary, endocrine, or renal disease that is uncontrolled or poorly controlled, any gastrointestinal illness (chronic reflux, inflammatory bowel disease, ulcer), any diabetes mellitus, and other such illnesses that can put a volunteer at increased risk. Exclusionary laboratory abnormalities include any abnormality that is grade 2 or above.
* Immunosuppressive illness or evidence of immunoglobulin A( IgA) deficiency (serum IgA < 7 mg/dL or below the limit of detection of assay). This includes any disease that requires immunosuppressive medication such corticosteroids, monoclonal antibodies that target key aspects of the immune system (e.g. rituximab or tumor necrosis factor (TNF) blockers, or any autoimmune disease).
* Positive serology results for HIV, HBsAg, or hepatitis C virus (HCV) antibodies, and confirmatory tests if appropriate.
* Positive urine toxicology screen for Amphetamines, Barbiturates, Benzodiazepines, cocaine metabolite, Methadone metabolite, Opiates, Oxycodone, and/or Phencyclidine.
* Significant abnormalities in screening laboratory hematology or serum chemistry, as determined by PI or PI in consultation with the research monitor and sponsor.
* Use of any medication known to affect immune function (e.g., regular systemic corticosteroids, monoclonal antibodies that target key aspects of the immune system (such as rituximab or tumor necrosis factor blockers); others [topical, intranasal and inhaled steroids will be permitted]) within 30 days preceding receipt of the investigational product or planned to be used during the active study period.
* Nursing or lactating on the day of admittance to the inpatient unit.
* Inability to tolerate 150 mL sodium bicarbonate buffer (based on requirement for frequent dosing).
* Recent vaccination (including licensed vaccines) or receipt of an investigational product (within 30 days before challenge through 30 days following the challenge dose).
* Prior history of C. difficile infection
* History of diarrhea in the 2 weeks prior to planned inpatient phase.
* Fewer than 3 stools per week or more than 3 stools per day as the usual frequency, or loose or liquid stools other than on an occasional basis.
* Regular use of laxatives or any agent that increases gastric pH (regular defined as at least weekly).
* Use of proton pump inhibitors, H2 blockers, or antacids within 48 hours of dosing.
* A fever (≥ 38.0°C) in the 2 weeks prior to time of challenge.
* Use of antibiotics during the 7 days before bacterial dosing or receipt of more than 2 courses of antibiotics over the two months prior to dosing.
* Blood donation within 30 days prior to the planned receipt of this investigational product.
* Lactose intolerance or allergy to milk or milk products.
* Personal or documented family history of Guillain-Barré syndrome or neuromuscular disease; or an inflammatory arthritis such as reactive arthritis, ankylosing spondylitis, or rheumatoid arthritis.
* Evidence of inflammatory arthritis on exam
* human leukocyte antigen B27(HLA B27) positive
* Allergy or prior intolerance to two or more of the following: fluoroquinolone, azithromycin, augmentin or cephalosporins.
* Have household contacts who are <2 years old or > 80 years old or infirm or immunocompromised.
* Employment as a healthcare worker with direct patient care, in a daycare center (for children or the elderly), or direct food handler; includes individuals who work directly with food in commercial establishments.
* History of microbiologically confirmed Campylobacter infection in the last 3 years.
* Serological immunological evidence of prior Campylobacter exposure as Campylobacter antigen-specific (GE) specific anti glycine extract serum IgA endpoint tier > 1:4,000.
* Occupation involving handling of Campylobacter currently, or in the past 3 years.
* Symptoms consistent with travelers' diarrhea concurrent with travel to countries where Campylobacter, Salmonella, Shigella, Typhoid or ETEC infection are endemic (most of the developing world) within 3 years prior to dosing, OR planned travel to endemic countries during the length of the study.
* Vaccination for or ingestion of Campylobacter, Cholera, Salmonella, Shigella, Typhoid or ETEC, within 5 years prior to dosing.
* Other dietary or environmental exposures that may place the participant at high risk for prior Campylobacter exposure (to be determined on a case by case basis by the PI).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2025-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar R Talaat, MD, Principal Investigator — Johns Hopkins Center for Immunization Research
Locations (1):
- Johns Hopkins University (Center for Immunization Research), Baltimore, Maryland, United States

REFERENCES:
- [Background] Scallan E, Hoekstra RM, Angulo FJ, Tauxe RV, Widdowson MA, Roy SL, Jones JL, Griffin PM. Foodborne illness acquired in the United States--major pathogens. Emerg Infect Dis. 2011 Jan;17(1):7-15. doi: 10.3201/eid1701.p11101. PMID 21192848
- [Background] Olson S, Hall A, Riddle MS, Porter CK. Travelers' diarrhea: update on the incidence, etiology and risk in military and similar populations - 1990-2005 versus 2005-2015, does a decade make a difference? Trop Dis Travel Med Vaccines. 2019 Jan 15;5:1. doi: 10.1186/s40794-018-0077-1. eCollection 2019. PMID 30675367
- [Background] Platts-Mills JA, Babji S, Bodhidatta L, Gratz J, Haque R, Havt A, McCormick BJ, McGrath M, Olortegui MP, Samie A, Shakoor S, Mondal D, Lima IF, Hariraju D, Rayamajhi BB, Qureshi S, Kabir F, Yori PP, Mufamadi B, Amour C, Carreon JD, Richard SA, Lang D, Bessong P, Mduma E, Ahmed T, Lima AA, Mason CJ, Zaidi AK, Bhutta ZA, Kosek M, Guerrant RL, Gottlieb M, Miller M, Kang G, Houpt ER; MAL-ED Network Investigators. Pathogen-specific burdens of community diarrhoea in developing countries: a multisite birth cohort study (MAL-ED). Lancet Glob Health. 2015 Sep;3(9):e564-75. doi: 10.1016/S2214-109X(15)00151-5. Epub 2015 Jul 19. PMID 26202075
- [Background] GBD 2016 Diarrhoeal Disease Collaborators. Estimates of the global, regional, and national morbidity, mortality, and aetiologies of diarrhoea in 195 countries: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Infect Dis. 2018 Nov;18(11):1211-1228. doi: 10.1016/S1473-3099(18)30362-1. Epub 2018 Sep 19. PMID 30243583
- [Background] Patrick ME, Henao OL, Robinson T, Geissler AL, Cronquist A, Hanna S, Hurd S, Medalla F, Pruckler J, Mahon BE. Features of illnesses caused by five species of Campylobacter, Foodborne Diseases Active Surveillance Network (FoodNet) - 2010-2015. Epidemiol Infect. 2018 Jan;146(1):1-10. doi: 10.1017/S0950268817002370. Epub 2017 Dec 14. PMID 29237513
- [Background] Connor BA, Riddle MS. Post-infectious sequelae of travelers' diarrhea. J Travel Med. 2013 Sep-Oct;20(5):303-12. doi: 10.1111/jtm.12049. Epub 2013 Jul 9. PMID 23992573
- [Background] Schwartz KL, Morris SK. Travel and the Spread of Drug-Resistant Bacteria. Curr Infect Dis Rep. 2018 Jun 29;20(9):29. doi: 10.1007/s11908-018-0634-9. PMID 29959541
- [Background] Novik V, Hofreuter D, Galan JE. Characterization of a Campylobacter jejuni VirK protein homolog as a novel virulence determinant. Infect Immun. 2009 Dec;77(12):5428-36. doi: 10.1128/IAI.00528-09. Epub 2009 Sep 21. PMID 19797067
- [Background] Parkhill J, Wren BW, Mungall K, Ketley JM, Churcher C, Basham D, Chillingworth T, Davies RM, Feltwell T, Holroyd S, Jagels K, Karlyshev AV, Moule S, Pallen MJ, Penn CW, Quail MA, Rajandream MA, Rutherford KM, van Vliet AH, Whitehead S, Barrell BG. The genome sequence of the food-borne pathogen Campylobacter jejuni reveals hypervariable sequences. Nature. 2000 Feb 10;403(6770):665-8. doi: 10.1038/35001088. PMID 10688204
- [Background] Karlyshev AV, Champion OL, Churcher C, Brisson JR, Jarrell HC, Gilbert M, Brochu D, St Michael F, Li J, Wakarchuk WW, Goodhead I, Sanders M, Stevens K, White B, Parkhill J, Wren BW, Szymanski CM. Analysis of Campylobacter jejuni capsular loci reveals multiple mechanisms for the generation of structural diversity and the ability to form complex heptoses. Mol Microbiol. 2005 Jan;55(1):90-103. doi: 10.1111/j.1365-2958.2004.04374.x. PMID 15612919
- [Background] Maue AC, Poly F, Guerry P. A capsule conjugate vaccine approach to prevent diarrheal disease caused by Campylobacter jejuni. Hum Vaccin Immunother. 2014;10(6):1499-504. doi: 10.4161/hv.27985. Epub 2014 Mar 14. PMID 24632556
- [Background] Pike BL, Guerry P, Poly F. Global Distribution of Campylobacter jejuni Penner Serotypes: A Systematic Review. PLoS One. 2013 Jun 27;8(6):e67375. doi: 10.1371/journal.pone.0067375. Print 2013. PMID 23826280
- [Background] Tacket CO, Losonsky G, Link H, Hoang Y, Guesry P, Hilpert H, Levine MM. Protection by milk immunoglobulin concentrate against oral challenge with enterotoxigenic Escherichia coli. N Engl J Med. 1988 May 12;318(19):1240-3. doi: 10.1056/NEJM198805123181904. PMID 3283555
- [Background] Tacket CO, Binion SB, Bostwick E, Losonsky G, Roy MJ, Edelman R. Efficacy of bovine milk immunoglobulin concentrate in preventing illness after Shigella flexneri challenge. Am J Trop Med Hyg. 1992 Sep;47(3):276-83. doi: 10.4269/ajtmh.1992.47.276. PMID 1524140
- [Background] Davidson GP, Whyte PB, Daniels E, Franklin K, Nunan H, McCloud PI, Moore AG, Moore DJ. Passive immunisation of children with bovine colostrum containing antibodies to human rotavirus. Lancet. 1989 Sep 23;2(8665):709-12. doi: 10.1016/s0140-6736(89)90771-x. PMID 2570959
- [Background] Savarino SJ, McKenzie R, Tribble DR, Porter CK, O'Dowd A, Cantrell JA, Sincock SA, Poole ST, DeNearing B, Woods CM, Kim H, Grahek SL, Brinkley C, Crabb JH, Bourgeois AL. Prophylactic Efficacy of Hyperimmune Bovine Colostral Antiadhesin Antibodies Against Enterotoxigenic Escherichia coli Diarrhea: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Trial. J Infect Dis. 2017 Jul 1;216(1):7-13. doi: 10.1093/infdis/jix144. PMID 28541500
- [Background] Savarino SJ, McKenzie R, Tribble DR, Porter CK, O'Dowd A, Sincock SA, Poole ST, DeNearing B, Woods CM, Kim H, Grahek SL, Brinkley C, Crabb JH, Bourgeois AL. Hyperimmune Bovine Colostral Anti-CS17 Antibodies Protect Against Enterotoxigenic Escherichia coli Diarrhea in a Randomized, Doubled-Blind, Placebo-Controlled Human Infection Model. J Infect Dis. 2019 Jul 2;220(3):505-513. doi: 10.1093/infdis/jiz135. PMID 30897198
- [Background] Freedman DJ, Tacket CO, Delehanty A, Maneval DR, Nataro J, Crabb JH. Milk immunoglobulin with specific activity against purified colonization factor antigens can protect against oral challenge with enterotoxigenic Escherichia coli. J Infect Dis. 1998 Mar;177(3):662-7. doi: 10.1086/514227. PMID 9498445
- [Background] Murray CJ, Vos T, Lozano R, Naghavi M, Flaxman AD, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gonzalez-Medina D, Gosselin R, Grainger R, Grant B, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Laden F, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Levinson D, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mock C, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiebe N, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, AlMazroa MA, Memish ZA. Disability-adjusted life years (DALYs) for 291 diseases and injuries in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2197-223. doi: 10.1016/S0140-6736(12)61689-4. PMID 23245608

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CampETEC HBC Group | Placebo ProMilk 85 Group
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CampETEC HBC Group | Placebo ProMilk 85 Group | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (5.1) | 36.5 (7.7) | 36.8 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 10 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black | 10 | 10 | 20
  White | 2 | 2 | 4
  Unknown | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 11 | 14 | 25
  Hispanic or Latino | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: The primary safety and tolerability outcome is the presence of CampETEC HBC associated adverse events during the study period. Safety of CampETEC HBC.
Time Frame: 28 days
Measure: Number (99% Confidence Interval); unit: events
Arm/Group | CampETEC HBC Group | Placebo ProMilk 85 Group
Number analyzed (Participants) | 13 | 14
events
  Abdominal distention | 1 [0.2 to 36.0] | 1 [0.2 to 33.9]
  Defaecation urgency | 0 [0.0 to 24.7] | 1 [0.2 to 33.9]
  Flatulence | 2 [1.9 to 45.4] | 2 [1.8 to 42.8]
  Gastrointestinal sounds abnormal | 0 [0.0 to 24.7] | 1 [0.2 to 33.9]
  Dizziness | 0 [0.0 to 24.7] | 1 [0.2 to 33.9]

2. Primary Outcome: Number of Participants With Campylobacteriosis Patterns
Description: The primary efficacy outcome is campylobacteriosis, defined as a clinical illness meeting at least one of the following patterns starting within 144 hours of challenge
  * Moderate diarrhea (4 to 5 loose/liquid stools or 401-800 grams in any 24 hour period) OR
  * Severe diarrhea (≥ 6 loose/liquid stools or > 800 grams in any 24 hour period) OR
  * Fever (present on at least 2 occasions, at least 20 minutes apart) without diarrhea, plus an associated symptom (nausea, vomiting, abdominal cramps, tenesmus, or dysentery (gross blood in ≥ 2 grade 3 - 5 stools with in any 24 hour period); with consideration of potential alternative diagnosis per clinical investigator based on illness time course and associated symptoms.
Time Frame: Within 144 hours of challenge
Measure: Count of Participants; unit: Participants
Arm/Group | CampETEC HBC Group | Placebo ProMilk 85 Group
Number analyzed (Participants) | 13 | 14
Participants
  Campylobacteriosis | 10 | 12
  Any Diarrhea | 10 | 11
  Mild Diarrhea | 0 | 0
  Moderate Diarrhea | 4 | 4
  Severe Diarrhea | 6 | 7
  Dysentery | 1 | 1
  Moderate/Severe Fever | 4 | 5
  Moderate/Severe Abdominal Pain/Cramps | 7 | 6
  Moderate/Severe Nausea | 3 | 3
  Moderate/Severe Vomiting | 0 | 0
  Moderate/Severe Anorexia | 4 | 3
  Early Antibiotic Treatment Required | 6 | 7
  IV Fluids Required | 1 | 3

ADVERSE EVENTS:
Time Frame: 28 days after Challenge
Description: CampETEC related Adverse Events
Arm/Group | CampETEC HBC Group | Placebo ProMilk 85 Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 10/13 | 11/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CampETEC HBC Group (N=13) | Placebo ProMilk 85 Group (N=14)
Abdominal distention (Gastrointestinal disorders) | 1 (1) | 1 (1) — CampETEC related AE
Defaecation Urgency (Gastrointestinal disorders) | 0 (0) | 1 (1) — CampETEC related AE
Flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2) — CampETEC related AE
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) — CampETEC related AE
Dizziness (General disorders) | 0 (0) | 1 (1) — CampETEC related AE
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Antibiotic related AE
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Antibiotic related AE
Vulvovaginal candidacies (Infections and infestations) | 1 (1) | 0 (0) — Antibiotic related AE
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Antibiotic related AE
Photophobia (Eye disorders) | 1 (1) | 0 (0) — Campylobacter Challenge related
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 5 (5) — Campylobacter Challenge related
Abdominal pain (Gastrointestinal disorders) | 10 (10) | 8 (8) — Campylobacter Challenge related
Abdominal rebound tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) — Campylobacter Challenge related
Abdominal tenderness (Gastrointestinal disorders) | 5 (5) | 2 (2) — Campylobacter Challenge related
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) — Campylobacter Challenge related
Defaecation urgency (Gastrointestinal disorders) | 5 (5) | 6 (6)
Flatulence (Gastrointestinal disorders) | 7 (7) | 6 (6) — Campylobacter Challenge related
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 2 (2) | 2 (2) — Campylobacter Challenge related
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) — Campylobacter Challenge related
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (3) — Campylobacter Challenge related
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) — Campylobacter Challenge related
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Campylobacter Challenge related
Chills (General disorders) | 7 (7) | 7 (7) — Campylobacter Challenge related
Malaise (General disorders) | 8 (8) | 8 (8) — Campylobacter Challenge related
Pyrexia (General disorders) | 6 (6) | 5 (5) — Campylobacter Challenge related
Dysentery (Infections and infestations) | 1 (1) | 1 (1) — Campylobacter Challenge related
Blood pressure decreased (Investigations) | 0 (0) | 1 (1) — Campylobacter Challenge related
Heart rate increased (Investigations) | 3 (3) | 4 (4) — Campylobacter Challenge related
Decreased Appetite (Metabolism and nutrition disorders) | 6 (6) | 7 (7) — Campylobacter Challenge related
Hypovolemia (General disorders) | 1 (1) | 1 (1) — Campylobacter Challenge related
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) — Campylobacter Challenge related
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Campylobacter Challenge related
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9) — Campylobacter Challenge related
Dizziness (Nervous system disorders) | 5 (5) | 3 (3) — Campylobacter Challenge related
Headache (Nervous system disorders) | 6 (6) | 11 (11) — Campylobacter Challenge related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/70/NCT06122870/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT06122870/ICF_001.pdf